CLINICAL TRIAL: NCT06497569
Title: Support Through Remote Observation and Nutrition Guidance Program for Individuals With Gastroesophageal Cancer (STRONG-GEC)
Brief Title: Support Through Remote Observation and Nutrition Guidance Program for Individuals With Gastroesophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-23230
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: GastroEsophageal Cancer
Keywords: Nutrition Support
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To reduce risk of bias, only assessors unaware of randomization status will be used to assess study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRONG Intervention (Experimental): Participants will receive an initial consultation and biweekly follow-up visits with a study dietitian for 90 days.
  During the follow-up visits, the study dietitian will review the dietary plan and goals, review the dietary food log, and discuss any challenges with dietary intake and recommendations for improving dietary intake.
  Participants will keep a daily diary of food intake with a Fitbit smartphone app and a Fitbit wearable device for 90 days, complete 6 questionnaires, and have the option to participate in a voluntary interview about the intervention.
  Interventions: Behavioral: Dietitian Consultation; Behavioral: Survey; Behavioral: Fitbit Data Collection; Behavioral: Social Determinants of Health Survey (SDOH)
- Usual Care Intervention (Active Comparator): Participants will be referred to a study dietitian based on their standard-care clinician's discretion, complete 6 questionnaires, and have the option to participate in a voluntary interview about the intervention.
  Interventions: Behavioral: Dietitian Consultation; Behavioral: Survey; Behavioral: Referral to Dietitian

INTERVENTIONS:
Behavioral: Dietitian Consultation — Participants will meet with a dietitian who will provide individualized nutrition counseling and dietary goals for calorie and protein intake.
  Bi-weekly, 30-minute dietitian telehealth visits will be conducted via ZOOM videoconferencing at the pre-intervention baseline visit, monthly during the intervention period (up to 90 days) and at the 4 and 6 month timepoints post-intervention.
Behavioral: Survey — Surveys will be conducted using the PG-SGA short form19-21 and a brief symptom assessment tool that captures additional nutrition-impact symptoms not captured by the PG-SGA (e.g., swallowing difficulty) measured by the FACT Esophageal and Gastric Cancer scales and the FAACT anorexia/cachexia scales 22,23 through REDCap.
  Surveys are completed at the pre-intervention baseline visit and monthly during the intervention period prior to the dietitian visits (up to 90 days), and at the 4 and 6 month timepoints post-intervention.
Behavioral: Fitbit Data Collection — Participants will log food intake while sharing their data with a dietitian during the 30-minute dietitian telehealth visits at the pre-intervention baseline visit, monthly during the intervention period (up to 90 days) and at the 4 and 6 month timepoints post-intervention.
  Arms: STRONG Intervention
Behavioral: Referral to Dietitian — Usual Care condition referral to a dietitian based on physician discretion.
  Arms: Usual Care Intervention
Behavioral: Social Determinants of Health Survey (SDOH) — Participants will complete a SDOH Survey that captures individual-level factors (insurance type, preferred language, educational attainment, annual household income, digital health literacy, financial toxicity, and self-reported barriers to care [e.g., transportation]) and structural-level factors (neighborhood disadvantage, rural residence).
  Digital health literacy will be measured using the validated eHEALS scale, an 8-item measure assessing confidence with finding, evaluating, and applying electronic information to inform health decision-making (score ≤ 30 indicates low literacy).
  Arms: STRONG Intervention

SUMMARY:
The purpose of this study is to determine how the STRONG intervention compares with usual care for reducing malnutrition among gastroesophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must have locally advanced or metastatic gastroesophageal cancer (GEC)
* Participants must plan to initiate chemotherapy and/or radiation therapy with a plan to have surgery or definitive treatment follow up at Moffitt
* Participants must be able to speak and read Spanish and/or English
* Participants must be able to provide informed consent

Exclusion Criteria:

* Participants have a documented or observable psychiatric or neurological disorder that would interfere with study participation (e.g. severe dementia)
* Use of feeding tubes at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate- Feasibility | Up to 48 Months
  The Study will be deemed feasible ≥ 50% of eligible patients are enrolled.
Retention Rate- Feasibility | Up to 90 Days
  The Study will be deemed feasible if ≥ 70% of participants enrolled at baseline are retained at the end of the intervention period.
Patient-reported outcome completion-Feasibility | Up to 6 Months
  The Study will be deemed feasible if ≥ 70% of participants enrolled submit 4 of the 6 study assessments.
Food Log Data Collection-Feasibility | Up to 6 Months
  The study will be deemed feasible if ≥ 70% of participants enrolled log food for greater than 80% of study days (72 out of 90).
Adherence to Dietitian Visits- Feasibility | Up to 6 Months
  The Study will be deemed feasible if ≥ 70% of participants enrolled attend 4 out of 6 dietitian visits.
Fidelity to Study Protocol- Feasibility | Up to 6 Months
  The Study will be deemed feasible if 20% of randomly audited dietitian visits have documented PG-SGA and calorie and protein goals
Patient Rating of MyPlate app-Feasibility | Up to 6 Months
  The Study will be deemed feasible if ≥ 70% of participants rate the MyPlate app as east-to use utilizing a validated usability scale (score ≥ 60).
Participant Satisfaction- Acceptability | Up to 6 Months
  Patient satisfaction with the intervention will be deemed acceptable if ≥ 70% of participants rate the intervention as satisfactory utilizing a validated 4 item scale (score range 0-20).
  A cutoff score of ≥ 12 based on prior studies to define intervention acceptability will be used.

SECONDARY OUTCOMES:
Malnutrition -Nutritional Status | Baseline, 3 Months, 6 Months
  Nutritional status will be measured using the Patient-Generated Subjective Global Assessment (PG-SGA) Short Form (score range: 0-35) and categorized based on a prior validation study (0-1 well nourished, 2-8 at-risk, ≥ 9 severely malnourished).
Malnutrition-Significant weight loss | Baseline, 3 Months, 6 Months
  Significant weight loss is defined as >5% and >10% of body weight. This will be calculated based on weight obtained during clinic visits.
Malnutrition - Low BMI | Baseline, 3 Months, 6 Months
  Low BMI will be defined as <20kg/m² for individuals <70 years old and <22kg/m2 for individuals ≥70 years old.
  This will be calculated based on weight and height measurements from clinic visits.
Malnutrition - Low Skeletal Muscle Mass | Baseline, 3 Months, 6 Months
  Low muscle mass will be estimated by calculating skeletal muscle index (SMI) from routinely collected CT scans at baseline, 3 months and 6 months (CT scans are conducted every 3 months). Low muscle mass will be defined as SMI ≤38.5 cm2 /m2 for females and SMI ≤52.4 cm2 /m2 for males.
Quality of Life Questionnaires | Baseline, 3 Months, 6 Months
  Quality of Life will be measured using the Functional Assessment of Cancer Therapy - General (FACT-G) Scale and the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) subscales.
  (FACT-G) and (FAACT) Questionnaires include questions about the participant's physical, social, emotional and functional well-being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher score indicates a better quality of life.
Treatment Adherence | Baseline, 3 Months, 6 Months
  Treatment Adherence will be measured by obtaining scheduling and electronic health record (EHR) data to estimate adherence to chemotherapy and/or radiation therapy.
  Comparison of will be made of planned vs. received chemotherapy and/or radiation regimens to define 1) treatment delay (yes/no); 2) dose reduction (yes/no); and 3) treatment discontinuation (yes/no). We will also document receipt of surgery (yes/no).
Progression Free Survival (PFS) | Up to 48 Months
  Progression Free Survival (PFS) status will be obtained from the cancer center registry to estimate overall survival (the time from random assignment to death from any cause) and progression-free survival (the time from random assignment to disease progression or death from any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Alishahi Tabriz, MD, PhD, MPH, Principal Investigator — Moffitt Cancer Center; Jose Pimiento, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — http://www.moffitt.org/clinical-trials-research/clinical-trials/